CLINICAL TRIAL: NCT03680274
Title: Lessening Organ Dysfunction With VITamin C (LOVIT)
Brief Title: Lessening Organ Dysfunction With VITamin C
Acronym: LOVIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Principal Investigator, François Lamontagne, Doctor, professor and researcher, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-31-2019-2945
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Sepsis; Vitamin C; Intensive Care Unit; COVID-19; Pandemic; Coronavirus
MeSH Terms: conditions — Sepsis; COVID-19; Coronavirus Infections | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Vitamin C: 50 mg/kg every 6 hours for 96 hours.
  Interventions: Drug: Vitamin C
- Control (Placebo Comparator): Dextrose 5% in water (D5W) or normal saline (0.9% NaCl) in a volume to match the vitamin C.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Vitamin C — Intravenous vitamin C administered in bolus doses of 50 mg/kg mixed in a 50-mL solution of either dextrose 5% in water (D5W) or normal saline (0.9% NaCl), during 30 to 60 minutes, every 6 hours for 96 hours (i.e. 200 mg/kg/day and 16 doses in total).
  Other Names: Ascorbic acid
  Arms: Vitamin C
Other: Control — Dextrose 5% in water (D5W) or normal saline (0.9% NaCl) in a volume to match the vitamin C.
  Arms: Control

SUMMARY:
LOVIT is a multicentre concealed-allocation parallel-group blinded randomized controlled trial to ascertain the effect of high-dose intravenous vitamin C compared to placebo on mortality or persistent organ dysfunction at 28 days in septic intensive care unit patients. Patients with COVID-19 are considered eligible for this study.

DETAILED DESCRIPTION:
Background. The burden of sepsis is increasing worldwide. It is the cause of 8 million global deaths each year. Currently, treatment options are limited to antimicrobials and supportive care such as intravenous fluids, vasopressors, mechanical ventilation, and renal replacement therapy. In the absence of effective therapies specifically targeting the dysregulated immune response, prolonged use of these life-sustaining therapies can be debilitating. A growing body of evidence suggesting that vitamin C, an inexpensive and readily available intervention, is potentially lifesaving in sepsis. Intravenous vitamin C may be the first therapy to mitigate the dysregulated cascade of events that leads to sepsis. If proven effective, vitamin C could be used worldwide and drastically change outcomes in high- and low-income settings alike.

Objectives. To determine whether intravenous vitamin C, compared to placebo, reduces mortality and morbidity in sepsis (induced by bacterial and viral pathogens (as COVID-19)), and compare clinical and biochemical measures of organ dysfunction, and health-related quality of life (HRQoL) at 6 months. To ascertain the volume of distribution, clearance, and plasma concentration over a course of 96 hours of intravenous vitamin C 50 mg/kg of weight every 6 hours or matching placebo (pharmacokinetic (PK) substudy).

Methods. Patients will be randomly assigned to vitamin C (intravenous, 50 mg/kg every 6h) or placebo (0.9% NaCl or dextrose 5% in water) for 96 hours. Study personnel at the clinical sites will document the composite of death or persistent organ dysfunction at day 28. Daily assessments will occur for organ function, on days 1, 3, 7 for inflammation, infection, and endothelial injury biomarkers, at baseline for vitamin C level, and at 6 months for mortality and HRQoL. The LOVIT Trial will be conducted in adult general Canadian and international intensive care units. For the PK substudy: Blood samples will be drawn around the 8th dose at time 0 and then after administration at times 1h, 2h, 4h and 6h (the 6h level will be immediately prior to the next dose). The PK substudy will be conducted with 100 participants in 3 of the 25 participating centers.

Relevance. In the context of increasing off-label use of vitamin C for sepsis and ongoing trials of vitamin C bundled with other pharmacological interventions, the LOVIT Trial will constitute a rigorous assessment of the effect of vitamin C monotherapy on patient-important outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the intensive care unit with proven or suspected infection as the main diagnosis;
2. Currently treated with a continuous IV infusion of vasopressors (norepinephrine, epinephrine, vasopressin, dopamine, phenylephrine).

Exclusion Criteria:

1. > 24 hours of intensive care unit admission;
2. Known Glucose-6-phosphate dehydrogenase (G6PD) deficiency;
3. Pregnancy;
4. Known allergy to vitamin C;
5. Known kidney stones within the past 1 year;
6. Received any intravenous vitamin C during this hospitalization unless incorporated in parenteral nutrition;
7. Expected death or withdrawal of life-sustaining treatments within 48 hours;
8. Previously enrolled in this study;
9. Previously enrolled in a trial with which co-enrolment is not allowed.

The LOVIT trial has broad eligibility criteria and includes patients with a primary diagnosis of sepsis of any cause (including sepsis caused by viral pathogens as COVID-19).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 872 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Number of deceased participants or with persistent organ dysfunction | Both assessed at 28 days
  Defined as death or dependency on mechanical ventilation, renal replacement, or vasopressors

SECONDARY OUTCOMES:
Number of participants with persistent organ dysfunction-free days in intensive care unit | Up to day 28
  Persistent organ dysfunction-free days in intensive care unit
Number of participants deceased at 6 months | 6 months
  Mortality at 6 months
Score of health related quality of life in 6-month survivors | 6 months
  Assessed by the questionnaire EuroQol-5D (EQ-5D-5L). The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Global tissue dysoxia | Days 1, 3, 7
  Assessed by serum lactate concentration
Organ function (including renal function) | Days 1, 2, 3, 4, 7, 10, 14, 28
  Assessed by the Sequential Organ Failure Assessment (SOFA) score. Used to track a person's status during the stay in an intensive care unit to determine the extent of a person's organ function or rate of failure. The score is based on 6 different sub-scores, one each for the respiratory (PaO2/FiO2 mmHg), cardiovascular (mean arterial pressure OR administration of vasopressors required), hepatic (liver bilirubin (mg/dl) [μmol/L]), coagulation (platelets×103/µl), renal (kidneys creatinine (mg/dl) [μmol/L] (or urine output)) and neurological (Glasgow coma scale). The sub-score of each system ranges from 0 (best) to +4 (worst).
Rate of inflammation | Days 1, 3, 7
  Assessed by interleukin-1 beta (IL-1ß), tumor necrosis factor-alpha (TNF-α), C-reactive protein (CRP).
Rate of infection | Days 1, 3, 7
  Assessed by procalcitonin (PCT)
Rate of endothelial injury | Days 1, 3, 7
  Assessed by thrombomodulin (TM) and angiopoietin-2 (ANG-2)
Occurrence of stage 3 acute kidney injury | Up to day 28
  Assessed by KDIGO (Kidney Disease: Improving Global Outcomes) criteria
Acute hemolysis | Up to day 28
  * clinician judgment of hemolysis, as recorded in the chart, OR
  * hemoglobin drop of at least 25 g/L within 24 hours of a dose of investigational product PLUS 2 of the following:
    * reticulocyte count >2 times upper limit of normal at clinical site lab;
    * haptoglobin < lower limit of normal at clinical site lab;
    * indirect (unconjugated) bilirubin >2 times upper limit of normal at clinical site lab;
    * Lactate dehydrogenase (LDH) >2 times upper limit of normal at clinical site lab.
  Severe hemolysis:
  - hemoglobin < 75 g/L AND at least 2 of the above criteria AND requires 2 units of packed red blood cells
Hypoglycemia | During the time participants receive the 16 doses of the investigational product and the 7 days following the last dose
  Core lab-validated glucose level of less than 3.8 mmol/L
Vitamin C volume of distribution | 8th dose of vitamin C at time 0 (immediately prior to the dose) and then after administration at times 1 hour, 2 hours, 4 hours and 6 hours (Pharmacokynetic substudy)
  Assessed by chromatography-tandem mass spectrometry
Vitamin C clearance | 8th dose of vitamin C at time 0 (immediately prior to the dose) and then after administration at times 1 hour, 2 hours, 4 hours and 6 hours (Pharmacokynetic substudy)
  Assessed by chromatography-tandem mass spectrometry
Vitamin C plasma concentration | 8th dose of vitamin C at time 0 (immediately prior to the dose) and then after administration at times 1 hour, 2 hours, 4 hours and 6 hours (Pharmacokynetic substudy)
  Assessed by chromatography-tandem mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: François Lamontagne, MD FRCPC MSc, Principal Investigator — Université de Sherbrooke and CIUSSS de l'Estrie - CHUS; Neill Adhikari, MDCM FRCPC MSc, Principal Investigator — Sunnybrook Health Sciences Centre, University of Toronto
Locations (1):
- Research Center of the CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data collected during the LOVIT trial will be shared with researchers who provide a detailed and methodologically sound proposal, with specific aims. Data sharing will be for the purposes of medical research, with specific data elements provided to answer the research questions in the proposal, and under the auspices of the consent under which the data were originally gathered.
Supporting Information: Study Protocol, SAP
Time Frame: Data availability will commence after the publication of the primary and secondary analyses, with no anticipated end date.
Access Criteria: Qualified researchers will need to sign a data sharing and access agreement and will need to confirm that data will only be used for the agreed upon purpose for which data access was granted. The decision to grant access will be made by the trial co-principal investigators, with involvement of the trial steering committee as needed. Proposals to access LOVIT data should be directed to the trial co-principal investigators via email: francois.lamontagne@usherbrooke.ca and neill.adhikari@utoronto.ca. Costs of preparing and providing partial datasets will be charged to requesting investigators.

REFERENCES:
- [Derived] Muller MM, Pinto R, Lamontagne F, Adhikari NKJ, Del Sorbo L; Lessening Organ Dysfunction With Vitamin C (LOVIT) Investigators. Vitamin C Does Not Affect Platelet Counts in Patients With Sepsis: A Post hoc Analysis of the Lessening Organ Dysfunction With Vitamin C Randomized Trial. Crit Care Explor. 2025 Sep 5;7(9):e1310. doi: 10.1097/CCE.0000000000001310. eCollection 2025 Sep. PMID 40927646
- [Derived] Rynne J, Mosavie M, Masse MH, Menard J, Battista MC, Maslove DM, Del Sorbo L, St-Arnaud C, DAragon F, Fox-Robichaud A, Charbonney E, Adhikari NKJ, Lamontagne F, Shankar-Hari M; LOVIT Investigators, the Canadian Critical Care Trials Group. Sepsis subtypes and differential treatment response to vitamin C: biological sub-study of the LOVIT trial. Intensive Care Med. 2025 Jan;51(1):82-93. doi: 10.1007/s00134-024-07733-9. Epub 2025 Jan 7. PMID 39774855
- [Derived] Lamontagne F, Masse MH, Menard J, Sprague S, Pinto R, Heyland DK, Cook DJ, Battista MC, Day AG, Guyatt GH, Kanji S, Parke R, McGuinness SP, Tirupakuzhi Vijayaraghavan BK, Annane D, Cohen D, Arabi YM, Bolduc B, Marinoff N, Rochwerg B, Millen T, Meade MO, Hand L, Watpool I, Porteous R, Young PJ, D'Aragon F, Belley-Cote EP, Carbonneau E, Clarke F, Maslove DM, Hunt M, Chasse M, Lebrasseur M, Lauzier F, Mehta S, Quiroz-Martinez H, Rewa OG, Charbonney E, Seely AJE, Kutsogiannis DJ, LeBlanc R, Mekontso-Dessap A, Mele TS, Turgeon AF, Wood G, Kohli SS, Shahin J, Twardowski P, Adhikari NKJ; LOVIT Investigators and the Canadian Critical Care Trials Group. Intravenous Vitamin C in Adults with Sepsis in the Intensive Care Unit. N Engl J Med. 2022 Jun 23;386(25):2387-2398. doi: 10.1056/NEJMoa2200644. Epub 2022 Jun 15. PMID 35704292
- [Derived] Lachance O, Goyer F, Adhikari NKJ, Masse MH, Bilodeau JF, Lamontagne F, Leclair MA. High-dose vitamin-C induced prolonged factitious hyperglycemia in a peritoneal dialysis patient: a case report. J Med Case Rep. 2021 May 21;15(1):297. doi: 10.1186/s13256-021-02869-4. PMID 34020705
- [Derived] Masse MH, Menard J, Sprague S, Battista MC, Cook DJ, Guyatt GH, Heyland DK, Kanji S, Pinto R, Day AG, Cohen D, Annane D, McGuinness S, Parke R, Carr A, Arabi Y, Vijayaraghavan BKT, D'Aragon F, Carbonneau E, Maslove D, Hunt M, Rochwerg B, Millen T, Chasse M, Lebrasseur M, Archambault P, Deblois E, Drouin C, Lellouche F, Lizotte P, Watpool I, Porteous R, Clarke F, Marinoff N, Belley-Cote E, Bolduc B, Walker S, Iazzetta J, Adhikari NKJ, Lamontagne F; Canadian Critical Care Trials Group. Lessening Organ dysfunction with VITamin C (LOVIT): protocol for a randomized controlled trial. Trials. 2020 Jan 8;21(1):42. doi: 10.1186/s13063-019-3834-1. PMID 31915072

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-01-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT03680274/SAP_000.pdf